CLINICAL TRIAL: NCT05289089
Title: The Well-being in IBS: Strengths and Happiness (WISH) Pilot Trial
Brief Title: Well-being in IBS: Strengths and Happiness (WISH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Elizabeth N. Madva, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P002996
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized trial comparing PP intervention versus wait list control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology Intervention Group (Experimental): Participants will complete 9 weekly phone sessions with a study trainer and positive psychology exercises between phone sessions. Study trainers will review the positive psychology exercises with the participant on the phone each week. Participants will receive this intervention in addition to their treatment as usual.
  Interventions: Behavioral: Positive Psychology Intervention
- Wait list Control Group (Active Comparator): After waiting for 9 weeks, participants will complete 9 weekly phone sessions with a study trainer and positive psychology exercises between phone sessions. Study trainers will review the positive psychology exercises with the participant on the phone each week. Participants will receive this intervention in addition to their treatment as usual.
  Interventions: Behavioral: Positive Psychology Intervention

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — Participants will receive a treatment manual. For each session, a PP exercise will be described in the manual, with instruments and space to write about the exercise and its effects. Participants will independently complete PP exercises between phone sessions and review them with their study trainer during phone sessions. A total of 9 sessions will be completed over the course of the program.

SUMMARY:
The purpose of this pilot study is to examine the feasibility, acceptability, and preliminary efficacy of a customized positive psychology (PP) intervention for patients with irritable bowel syndrome (IBS) compared to a wait list control group.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS), a disorder of gut-brain interaction (DGBI; formerly known as functional gastrointestinal disorder) is characterized by abdominal pain and altered bowel habits, and conceptualized as resulting from complex interactions between biological, psychological, and social factors.

The treatment approach for IBS is multifaceted and focused on symptom reduction rather than cure. For mild or infrequent symptoms, lifestyle modification (e.g., diet and exercise), reassurance, and education about the disorder can at times be sufficient. For moderate to severe symptoms, a combination of pharmacotherapy and behavioral health interventions is often required. A growing body of evidence supports the use of behavioral health interventions to target the gut-brain axis in DGBI - aptly referred to as brain-gut behavior therapies (BGBT). Though highly effective, existing BGBT for IBS face important limitations including scalability and acceptability. There is also limited focus among existing BGBT on the promotion of positive psychological (PP) constructs (e.g., optimism), which are deficient in IBS, associated with fewer IBS symptoms, and associated with lower levels of distress in both clinical and non-clinical populations.

PP interventions have successfully been implemented in a variety of other chronic medical conditions to improve well-being, health-related quality of life, and health behavior engagement. PP interventions are highly acceptable and easily delivered remotely without extensive specialized training, which increases their scalability and reach.

As such, the investigators plan to do the following in this project:

1. Examine the feasibility and acceptability of a 9-week, telephone-delivered PP intervention adapted to the IBS population
2. Explore the impact of the PP intervention on psychological, behavioral, and health-related outcomes, compared to a wait list control group.

ELIGIBILITY:
Inclusion Criteria:

* IBS Diagnosis: Adult patients with an IBS diagnosis documented by the patient's primary care or GI clinician and meeting standardized ROME IV diagnostic criteria.
* Language and communication: English fluency and access to a telephone.

Exclusion Criteria:

* Severe psychiatric illness: Current manic episode, psychosis, or active substance use disorder diagnosed via the Mini International Neuropsychiatric Interview (MINI).
* Cognitive impairment: Assessed using a six-item cognitive screen developed for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Proportion of PP Sessions Completed by Participants | 9 weeks
  Measured by proportion of PP sessions completed by participants in each group.

SECONDARY OUTCOMES:
Ease of PP Exercises | Weeks 1-9
  Participants will provide ratings of ease after each PP exercise, measured on a 10-point Likert scale (0=very difficult, 10=very easy). Weekly ratings will be averaged to provide an overall ease of the exercises.
Utility of PP exercises | Weeks 1-9
  Participants will provide ratings of utility after each PP exercise, measured on a 10-point Likert scale (0=not at all helpful; 10=very helpful). Weekly utility ratings will be averaged to provide an overall utility score of the exercises.
Change in Positive Affect | Change in score from Baseline to 9 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Optimism | Change in score from Baseline to 9 weeks
  Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of optimism. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Depression | Change in score from Baseline to 9 weeks
  The Hospital Anxiety and Depression Scale (HADS)-depression subscale will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Anxiety | Change in score from Baseline to 9 weeks
  The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale will be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Gastrointestinal (GI) symptom specific anxiety | Change in score from Baseline to 9 weeks
  Measured by the Visceral Sensitivity Index (VSI) score, a validated self-report measure of anxiety specific to visceral sensations (Range: 0-75). Higher scores indicate higher levels of GI-specific anxiety. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Ability to Bounce Back from Stress | Change in score from Baseline to 9 weeks
  Measured by the Brief Resilience Scale (BRS) (Range: 6-30), a reliable 6-item measure of the ability to "bounce back" or recover from stress. Higher scores reflect greater bounce back resilience. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Ability to Cope with Stress and Adversity | Change in score from Baseline to 9 weeks
  Measured by the 25-item Connor-Davidson Resilience Scale (CD-RISC) (Range: 0-100), a reliable and validated measure of resilience, defined as the ability to cope with stress and adversity. Higher scores reflect greater resilience. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Response to Pain | Change in score from Baseline to 9 weeks
  Measured by the Pain Catastrophizing Scale (PCS), a widely used tool to assess cognitive and affective responses to pain (Range: 0-52). Higher scores indicate higher levels of pain-related anxiety. Change will be calculated by subtracting the scores at baseline from the scores at 9 weeks.
Change in Perceived Stress | Change in score from Baseline to 9 weeks
  Measured by the Perceived Stress Scale (PSS) (Range: 0-40). Higher scores indicate higher perceived stress. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in IBS Health-related Quality of Life | Change in score from Baseline to 9 weeks
  Measured by the IBS Quality of Life (IBS-QOL) score (Range: 0-100), a validated disease-specific instrument measuring quality of life. Higher scores indicate better IBS-specific quality of life. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in IBS Symptom Severity | Change in score from Baseline to 9 weeks
  Measured by the IBS symptom severity score (IBS-SSS) score (Range: 0-500), a validated disease-specific instrument measuring symptom severity. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Self-Reported Physical Activity | Change in score from Baseline to 9 weeks
  Measured by the self-report International Physical Activity Questionnaire (IPAQ). This measure assesses the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Adherence to a Physician-Recommended Diet | Change in score from Baseline to 9 weeks
  Measured with a single question inquiring if the participant followed the diet with possible responses including: never, a quarter of the time, half of the time, three-quarters of the time, or always. A score of 0-4 (0=never, 4=always) will be applied. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Adherence to Medications | Change in score from Baseline to 9 weeks
  Measured with a 3-item questionnaire from the Heart and Soul study. Participants will be categorized as adherent (>75% of the time) versus non-adherent (<75% of the time), and this will be compared between baseline and 9 weeks.
Change in Avoidant and Restrictive Food Intake Disorder Symptoms | Change in score from Baseline to 9 weeks
  Measured by the Nine Item Avoidant/Restrictive Food Intake Disorder screen (NIAS) (Range: 0-45), a validated tool to assess avoidant/restrictive eating patterns. Higher scores indicate higher levels of avoidant/restrictive eating patterns. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in Eating Behaviors | Change in score from Baseline to 9 weeks
  Measured by the Eating Disorder Examination Questionnaire 8 (EDE-Q8) (Range: 0-6), an 8-item questionnaire that assesses eating disorder symptoms over the past 28 days. Higher scores indicate higher levels of eating disordered symptoms. Change will be calculated by subtracting the score at baseline from the score at 9 weeks.
Change in IBS diagnostic criteria | Change in score from Baseline to 9 weeks
  Measured by the Rome IV Diagnostic Questionnaire - Irritable Bowel Syndrome (IBS) Module. This questionnaire provides inclusion criteria for IBS for clinical research studies. To meet criteria for IBS, participants must have the following for the past 3 months: (1) recurrent abdominal pain at least weekly; (2) pain associated with 2 or more of the following criteria: (a) related to defecation at least 30% of occasions; (b) associated with change in stool frequency at least 30% of occasions; (c) associated with change in stool form at least 30% of occasions; and (3) symptom onset at least 6 months prior to diagnosis.
Immediate Impact of the Exercises: Change in Optimism Ratings | Weeks 1-9
  Participants will provide ratings of optimism before and after each positive psychology exercise, measured on a 10-point Likert scale (0-10). Higher scores indicate higher levels of optimism.
Immediate Impact of the Exercises: Change in Happiness Ratings | Weeks 1-9
  Participants will provide ratings of happiness before and after each positive psychology exercise, measured on a 10-point Likert scale (0-10). Higher scores indicate higher levels of happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Madva, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No